CLINICAL TRIAL: NCT04941833
Title: The Use of Oral Desogestrel for the Preoperative Treatment of Endometrioma Compared With Placebo : A Randomized Controlled Trial Evaluation of the Effect on Cyst Diameter and Associated Pain
Brief Title: Desogestrel for the Preoperative Treatment of Endometrioma Compared With Placebo
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 147/2564
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Endometrioma
MeSH Terms: conditions — Endometriosis | interventions — Desogestrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desogestrel group (Experimental): Desogestrel group
  Interventions: Drug: Desogestrel Oral Tablet
- Control group (Placebo Comparator): Placebo
  Interventions: Drug: Desogestrel Oral Tablet

INTERVENTIONS:
Drug: Desogestrel Oral Tablet — Cerazette is the brand name of the desogestrel which contain of 0.075 mg of desogestrel
  Other Names: Cerazette

SUMMARY:
Use of the oral desogestrel compared with placebo for preoperative treatment of endometrioma in the patient who underwent to surgery in next 3 months The result will be evaluated on cyst diameter, the associated pain and side effect of the oral desogestrel.

DETAILED DESCRIPTION:
Use of the oral desogestrel compared with placebo for preoperative treatment of endometrioma in the patient who underwent to surgery in next 3 months in Rajvithi hospital Patient will randomized in 2 group : Desogestrel and placebo After 1 months and 3 months the patient have to come to hospital to evaluate the result of study The result will be evaluated on cyst diameter, the associated pain and side effect of the oral desogestrel.

ELIGIBILITY:
Inclusion Criteria:

* Thai female and foreigner who can understand Thai language
* Age 15-49 years
* Diagnose as endometrioma sized more than 3 cm
* Underwent to surgery in next 13 weeks

Exclusion Criteria:

* History of endometriosis
* Pregnancy woman
* Contraindication for desogestrel : History of thrombotic event, Autoimmune disease,gestational trophoblastic disease
* Ovarian endometrioma with complications : Ruptured, twisted
* Contraindications for NSAIDs : Peptic ulcer, thrombocytopenia, liver disease
* History of hormonal treatment for endometrioma : DMPA,OCP, GNRH agonist/antoginist

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Cyst diameter | 3 months after drug given
  Cyst diameter is calculated by transvaginal ultrasound with calculated in the diameter of endometrimas (cm)

SECONDARY OUTCOMES:
Associated pain | 3 months after drug given
  Associated pain is measured by the visual analog score. The patients will record the score on the book everytimes when they have pain

OTHER OUTCOMES:
Effect of the drug in the study | 3 months after drug given
  Effect of the oral desogestrel and placebo such as spotting, weight gain, wood swing

CONTACTS AND LOCATIONS:
Overall Officials: Ratchadaporn Roekyindee, MD, Study Director — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muzii L, Galati G, Di Tucci C, Di Feliciantonio M, Perniola G, Di Donato V, Benedetti Panici P, Vignali M. Medical treatment of ovarian endometriomas: a prospective evaluation of the effect of dienogest on ovarian reserve, cyst diameter, and associated pain. Gynecol Endocrinol. 2020 Jan;36(1):81-83. doi: 10.1080/09513590.2019.1640199. Epub 2019 Jul 14. PMID 31304853
- [Background] Cucinella G, Granese R, Calagna G, Svelato A, Saitta S, Tonni G, De Franciscis P, Colacurci N, Perino A. Oral contraceptives in the prevention of endometrioma recurrence: does the different progestins used make a difference? Arch Gynecol Obstet. 2013 Oct;288(4):821-7. doi: 10.1007/s00404-013-2841-9. Epub 2013 Apr 12. PMID 23580011
- [Background] Taniguchi F, Enatsu A, Ota I, Toda T, Arata K, Harada T. Effects of low dose oral contraceptive pill containing drospirenone/ethinylestradiol in patients with endometrioma. Eur J Obstet Gynecol Reprod Biol. 2015 Aug;191:116-20. doi: 10.1016/j.ejogrb.2015.06.006. Epub 2015 Jun 16. PMID 26115056
- [Background] Razzi S, Luisi S, Ferretti C, Calonaci F, Gabbanini M, Mazzini M, Petraglia F. Use of a progestogen only preparation containing desogestrel in the treatment of recurrent pelvic pain after conservative surgery for endometriosis. Eur J Obstet Gynecol Reprod Biol. 2007 Dec;135(2):188-90. doi: 10.1016/j.ejogrb.2006.08.002. Epub 2006 Sep 11. PMID 16963174